CLINICAL TRIAL: NCT00688532
Title: A Pharmacoepidemiological Study on the Association Between Bicalutamide Treated Prostate Cancer and Risk of Coronary Heart Disease (CHD) and Heart Failure (HF) in the General Practice Research Database (GPRD)
Brief Title: Study of Coronary Heart Disease (CHD) & Heart Failure (HF) Risk in Prostate Cancer Patients, Taking Casodex or Not
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D6874C00008
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; pharmacoepidemiology study
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Prostate cancer patients treated with bicalutamide or not
- 2: General population cohort

SUMMARY:
A retrospective cohort study performed in the GPRD,UK. All patients with incident prostate cancer identified between 1 Jan 1999 and 31 Dec 2005 and a frequency-matched cohort of the general population will be followed- up for two outcomes; CHD including acute myocardial infarction or death from coronary heart disease and HF until Dec 31, 2006. Outcomes will be validated through requests to primary care physicians. Incidence rate´ratios of CHD and HF in the two cohorts will be calculated. In the cohort of prostate cancer the relative risk of CHD and HF associated with the use of bicalutamide compared to non-use will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* At least two years enrollment with the general practitioner

Exclusion Criteria:

* Patients with cancer before start date of the study

Ages: 50 Years to 84 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GPRD containing computerized information entered by general practitioners in the UK
Sampling Method: Probability Sample
Enrollment: 5103 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Coronary heart disease including acute myocardial infarction and death from CHD | From study start 1 Jan 1999 through 31December 2006
Heart Failure | From study start 1 Jan 1999 through 31December 2006

CONTACTS AND LOCATIONS:
Overall Officials: LA García Rodríguez, MD, Principal Investigator — CEIFE (Centro Español de Investigación Farmacoepidemiológica -Spanish Centre for Pharmacoepidemiologic Research) Almirante